CLINICAL TRIAL: NCT01397851
Title: Stimulating Private Sector Malaria Control: The Outgrower Opportunity
Brief Title: Stimulating Private Sector Malaria Control
Acronym: Outgrowers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Principal Investigator, Elizabeth Trias, Principal Investigator, PATH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PATH Outgrowers
Record Dates: First submitted 2011-06-21; First posted 2011-07-20 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment: Insecticide-treated net (Experimental): Smallholder farmers in the treatment group are informed that they won a raffle, and receive a free insecticide-treated net
  Interventions: Device: Insecticide-treated net (BASF Incerceptor)
- Control (No Intervention): Smallholder farmers in the control group are informed that they had a chance to win an insecticide-treated mosquito net in a raffle, but did not end up winning

INTERVENTIONS:
Device: Insecticide-treated net (BASF Incerceptor) — One per farmer, once during the 2010-2011 season
  Arms: Treatment: Insecticide-treated net

SUMMARY:
Preliminary evidence from ongoing research provides strong indications that protecting farmers from malaria would be profitable for outgrowing agribusinesses in sub-Saharan Africa. The study team invests in experimental research to investigate this conjecture in more detail.

DETAILED DESCRIPTION:
The study evaluates whether the sourcing of insecticide-treated nets and their distribution to smallholder farmers for free would be a profitable investment for a cotton outgrowing agribusiness in Zambia.

The study therefore carries out a major net distribution through the existing distribution channels of a cotton outgrowing agribusiness, evaluates the impact of this distribution on smallholder cotton yields, and values the profitability implications for the outgrowing agribusiness.

ELIGIBILITY:
Inclusion Criteria:

* Farmers who contracted with the participating cotton outgrowing company in the 2010-2011 season

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81597 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Malaria Control Centre, Lusaka, Zambia

REFERENCES:
- See also: status update as of 2 April 2013 — http://www.openscienceframework.org/project/vdS5m/node/253iA/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Treatment
Started | 41634 | 39963
Completed | 41555 | 39917
Not Completed | 79 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment: Insecticide-treated Net | Control | Total
Number analyzed (Participants) | 39963 | 41634 | 81597
Age, Continuous [Mean (Standard Deviation)] | NA (NA) — not collected | NA (NA) — not collected | NA (NA) — not collected
Sex/Gender, Customized [Number]
  Female | NA — not collected | NA — not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — not collected | NA — not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  Zambia | 39963 | 41634 | 81597

OUTCOME MEASURES:

1. Primary Outcome: Cotton Yields
Description: Farmer's cotton yields (kg delivered per household), as defined in the routine data collection system of the participating cotton outgrowing agribusiness
Time Frame: 2010-2011 season (up to 1 year)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Treatment: Insecticide-treated Net | Control
Number analyzed (Participants) | 39917 | 41555
kg | 544 (11) | 548 (11)

2. Secondary Outcome: Contract Defaults
Description: Defaults on input loans, as defined in the routine data collection system of the participating cotton outgrowing agribusiness. Odds ratios calculated in accordance with NIH guidance: http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2938757/
Time Frame: 2010-2011 season (up to 1 year)
Measure: Number; unit: odds ratio
Arm/Group | Treatment: Insecticide-treated Net | Control
Number analyzed (Participants) | 39917 | 41555
odds ratio | 0.887 | 1.127

3. Secondary Outcome: Increase in Maize Productivity
Description: Increase in self-reported maize productivity (yield on maize plots divided by size of maize plots), collected through validation survey; calculated as maize productivity 2010-11 minus maize productivity 2009-10, measured in bags (ordinarily 50kg bags; however, kg measure not specified)
Time Frame: 2009-2010 and 2010-2011 seasons (up to 2 years)
Population: Subset of study population selected for validation survey
Measure: Mean (Standard Error); unit: bags (not further specified)
Arm/Group | Treatment: Insecticide-treated Net | Control
Number analyzed (Participants) | 720 | 720
bags (not further specified) | 55 (6) | 59 (6)

4. Secondary Outcome: Self-reported Malaria Prevalence
Description: Over two weeks before interview, collected through validation survey. Odds ratio calculated in accordance with NIH guidance http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2938757/
Time Frame: 2010-2011 season (up to 1 year)
Population: Subset of study population selected for validation survey
Measure: Number; unit: odds ratio
Arm/Group | Treatment: Insecticide-treated Net | Control
Number analyzed (Participants) | 720 | 720
odds ratio | 0.58 | 1.72

ADVERSE EVENTS:
Description: No participants were deemed at risk of adverse events; no data on adverse events was collected
Arm/Group | Treatment: Insecticide-treated Net | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No